CLINICAL TRIAL: NCT03018041
Title: The Long-term Effect of Marine n-3 Polyunsaturated Fatty Acid Supplementation on Glomerular Filtration Rate and Development of Fibrosis in the Renal Allograft: a Randomized Double Blind Placebo Controlled Intervention Study
Brief Title: The Long-term Effect of Marine Omega-3 Fatty Acid Supplementation in Renal Transplantation
Acronym: EMiRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joe Chan (Other)
Collaborators: University of Oslo (Other); Rikshospitalet University Hospital (Other); Ullevaal University Hospital (Other); Drammen sykehus (Other); Elverum Hospital (Unknown); South-Eastern Norway Regional Health Authority (Other); Aalborg University Hospital (Other); Pronova BioPharma (Industry); Haukeland University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor-Investigator, Joe Chan, MD, PhD, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1652 (REK); 2016-003537-18 (EudraCT Number)
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Renal transplantation; Omega-3 fatty acids; Marine n-3 fatty acids; Fatty acids; Inflammation; Interstitial fibrosis; Glomerular filtration rate; Renal function; Allograft function; Proteinuria; Blood pressure; Heart rate variability; Lipids; Blood glucose; Body mass index; Fatty acid composition; Gas chromatography; Interventional study; Allograft biopsy; Kidney biopsy
MeSH Terms: conditions — Inflammation; Pulmonary Fibrosis; Proteinuria | interventions — Omacor; Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marine n-3 PUFAs (Experimental): 3 capsules of Omacor 1000 mg daily, corresponding to a dose of 2.5 g / day of marine n-3 PUFAs (EPA plus DHA).
  Interventions: Drug: Omacor
- Placebo (Placebo Comparator): Corresponding placebo oral capsules with olive oil, three capsules daily.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Omacor — As described in "Arms".
  Other Names: Omega-3 fatty acids; EPA; DHA; Marine n-3 polyunsaturated fatty acids
  Arms: Marine n-3 PUFAs
Drug: Placebo Oral Capsule — As described in "Arms".
  Other Names: Olive oil
  Arms: Placebo

SUMMARY:
This is a long-term intervention study on the effects of marine n-3 PUFAs in renal transplantation. Our hypothesis is that patients treated with marine n-3 PUFA supplementation will have less decline in kidney transplant function compared to patients treated with placebo.

DETAILED DESCRIPTION:
The study is designed as a randomized, double blind, placebo controlled, multi-center trial of 174 renal transplant recipients. Patients will be randomized to oral supplementation of marine n-3 PUFA 2.5 g / day or control in a 1:1 fashion.

The primary endpoint is change in estimated glomerular filtration rate after 156 weeks in the treatment group compared with the control group. Secondary endpoints include the following variables: proteinuria, plasma inflammatory biomarkers, blood pressure, resting heart rate, fasting serum glucose / HbA1c, lipid and lipoprotein concentrations, number of graft rejections and graft losses, and number of cardiovascular events and deaths.

Patients from Akershus University Hospital will also participate in a sub-study, where renal graft biopsies will be performed to assess the degree of fibrosis and chronic allograft damage index (CADI) and markers of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients over 18 years of age.
* Stable renal graft function, defined as eGFR >30 ml/min at the last 2 visits.
* 6-60 months post-transplantation at randomization.
* Signed informed consent.

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the last dose of study drug.
* Women who are pregnant or breastfeeding.
* Patients who participate in a clinical trial with other investigational drugs.
* Patients with a history of an allergic reaction or significant sensitivity to fish, seafood and the study drug Omacor or drugs or dietary supplements similar to the study drug.
* Any reason why, in the opinion of the Principal Investigator, the patient should not participate - E.g. history of repeated non-adherence to prescribed treatment, repeated non-attendance to clinic visits, cognitive impairment that prevents understanding the nature of this study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 156 weeks
  Estimated by CKD-EPI equation

SECONDARY OUTCOMES:
Proteinuria | 156 weeks
  ACR and FE-protein
Plasma fatty acid levels | 156 weeks
  measured by gas chromatography
Plasma inflammatory biomarkers | 156 weeks
Blood pressure | 156 weeks
Resting heart rate | 156 weeks
Fasting serum glucose / HbA1c | 156 weeks
Lipid and lipoprotein concentrations | 156 weeks
Body mass index | 156 weeks
Heart rate variability | 156 weeks
  Sub-study, participants from Akershus University Hospital only
The degree of fibrosis and chronic allograft damage index (CADI) in renal cortical tissue | 156 weeks
  Sub-study, participants from Akershus University Hospital only
Markers of fibrosis in renal cortical tissue | 156 weeks
  Sub-study, participants from Akershus University Hospital only
Fatty acid levels in renal cortical tissue | 156 weeks
  Sub-study, participants from Akershus University Hospital only

OTHER OUTCOMES:
Adverse events | 156 weeks
  Incl. number of graft rejections and losses, cardiovascular events and deaths
Adverse reactions | 156 weeks

CONTACTS AND LOCATIONS:
Overall Officials: My Svensson, MD, PhD, Study Director — University Hospital, Akershus; Ivar Anders Eide, MD, PhD, Study Chair — University Hospital, Akershus; Branimir Draganov, MD, Study Chair — Ullevaal University Hospital; Joe Chan, MD, Principal Investigator — University Hospital, Akershus; Morten Reier-Nilsen, MD, Principal Investigator — Drammen sykehus; Tone Granseth, MD, Principal Investigator — Elverum Hospital; Nanna von der Lippe, MD, PhD, Principal Investigator — Ullevaal University Hospital; Bård Endre Waldum-Grevbo, MD, PhD, Principal Investigator — Ullevaal University Hospital; Per Olav Rui, MD, Principal Investigator — Haukeland University Hospital; Toralf Melsom, MD, PhD, Principal Investigator — University Hospital of North Norway; Renathe Rismo, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (6):
- Norway (6):
  - Akershus University Hospital, Lørenskog, Akershus
  - Drammen Hospital, Drammen, Buskerud
  - Elverum Hospital, Elverum, Hedmark
  - Ullevaal University Hospital, Oslo, Oslo County
  - Haukeland University Hospital, Bergen
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No